CLINICAL TRIAL: NCT07022405
Title: Stratified Pharmacological Approaches for Regulating Circuit-Level Effects Study
Brief Title: Stratified Pharmacological Approaches for Regulating Circuit-Level Effects
Acronym: SPARCLE
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Leanne Williams, Professor of Psychiatry and Behavioral Sciences, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 80975; 5U01MH136062-02 (NIH)
Record Dates: First submitted 2025-06-06; First posted 2025-06-15 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Depression - Major Depressive Disorder
MeSH Terms: interventions — Pramipexole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pramipexole Treatment Arm (Experimental): The investigators will ask eligible participants to attend up to 2 in-person testing visits and commit to 10 weeks of treatment and remote participation.
  The in-person testing visit at the beginning of the study lasts up to 4 hours. During this visit participants will undergo a non-invasive functional magnetic resonance imaging (fMRI) brain scan, complete game-like tasks in the scanner, and answer questions regarding emotional health.
  Treatment involves an 8-week course of pramipexole and followed by a 2-week down titration and follow up. During this 10-week period, participants will meet remotely with a study coordinator or study clinician each week to answer questions about medication side effects and emotional health and to complete online surveys to monitor mood.
  Interventions: Drug: Pramipexole Immediate Release

INTERVENTIONS:
Drug: Pramipexole Immediate Release — The intervention involves taking pramipexole immediate release (IR) for 8 weeks followed by 2 weeks of down titration and follow up.

SUMMARY:
This research study aims to understand how people with depression respond to the medication pramipexole and to determine whether clinical response differs depending on the function of specific circuits in the brain. The investigators hope to learn which circuits are involved in depression and how these circuits interact with pramipexole to affect mood, behavior, and cognition.

Eligible participants will undergo an 8-week treatment course of pramipexole followed by a 2-week down taper and follow up. The ultimate goal is to offer people experiencing depression a medication that is alternative to ones that may not have worked in the past and to apply the knowledge the investigators gain from investigating the brain circuits involved in depression to help personalize treatment.

The investigators invite anyone who has recently experienced symptoms of depression to participate. A prior diagnosis of depression is not required.

DETAILED DESCRIPTION:
Participants will be asked to attend up to two in-person testing visits and commit to 10 weeks of treatment and remote participation.

The in-person testing visit at the beginning of the study lasts up to 4 hours. During this visit participants will undergo a non-invasive functional magnetic resonance imaging (fMRI) brain scan, complete game-like tasks in the scanner, and answer questions regarding emotional health.

Treatment involves an 8-week course of pramipexole and followed by a 2-week down taper and follow-up. During this 10-week period, participants will meet remotely with a study coordinator or study clinician each week to answer questions about medication side effects and emotional health and to complete online surveys to monitor mood.

Sign up online or contact the investigators to learn more about participating in this study.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old (inclusive)
* Fluent and literate in English, with non-impaired intellectual abilities to ensure adequate comprehension of the task instructions.
* Willing to provide written, informed consent.
* Functional magnetic resonance imaging (fMRI) scanning eligibility. All participants will need to successfully complete the screening forms at the Stanford Center for Cognitive and Neurobiological Imaging (CNI).
* Patient Health Questionnaire-8 (PHQ-8) >/= 10
* Meet the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) diagnostic criteria for current or recurrent nonpsychotic Major Depressive Disorder (MDD) established by the Mini International Neuropsychiatric Interview (MINI)

Exclusion Criteria:

* Suicidality with active plan or as determined clinician judgment
* Current or lifetime history of medical illness or brain injury that may interfere with assessments as determined by clinician judgment
* Severe impediment to vision, hearing, and/or hand movement likely to interfere with ability to complete the assessments, or is unable and/or unlikely to follow the study protocols as determined by clinician judgment
* Pregnant, breastfeeding or unwilling or unable to use adequate birth control throughout the study
* History of non-responsive depression to dopamine agonists
* Any contraindication to being scanned in the 3.0T fMRI scanner, such as a cardiac pacemaker or implanted device that has not been cleared for scanning
* Previous or current DSM-5 bipolar disorder (I, II, not otherwise specified), schizophrenia spectrum or other psychotic disorders, or psychosis or as determined by clinician judgment
* Previous or current diagnosis of Attention-Deficit/Hyperactivity Disorder (ADHD)
* Meeting DSM-5 criteria for current Obsessive-Compulsive Disorder (OCD) or eating disorder
* Meeting DSM-5 criteria for alcohol use disorder or substance use disorder within the last 12 months
* Clinically significant presence/history of impulsive-compulsive behaviors or control disorder including but not limited to gambling disorder within the last 12 months.
* Current use or use of psychotropic medication within the past month. (If the participant's usual treating clinician agrees with discontinuing the medication, participants may enroll after tapering off the medication under the supervision of either their usual clinician or the study clinician. A washout period of 5 half-lives-or a different duration as determined by the study clinician-must be completed before the first scan.)
* Concurrent participation in other intervention or treatment studies
* Not having a current primary care or psychiatric provider (seen within the past year)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2030-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
QIDS-SR: Quick Inventory of Depressive Symptomatology Self-Report | 8 weeks
  The QIDS-SR (Quick Inventory of Depressive Symptomatology - Self-Report) is a self-report questionnaire designed to assess the severity of depressive symptoms over the past seven days. It includes 16 items that evaluate 9 symptom domains corresponding to the Diagnostic and Statistical Manual of Mental Disorders (DSM) criteria for major depressive disorder: sad mood, concentration difficulties, self-criticism or guilt, suicidal ideation, loss of interest, low energy or fatigue, sleep disturbances, changes in appetite or weight, and psychomotor agitation or retardation. Each domain is rated on a scale from 0 to 3, with total scores ranging from 0 to 27. Scores are interpreted as follows: 0-5 indicates no depression, 6-10 mild, 11-15 moderate, 16-20 severe, and 21-27 very severe depression. It is brief, taking approximately 5 to 10 minutes to complete.
MASQ-30: Mood Anxiety Symptom Questionnaire | 8 weeks
  The MASQ-30 (Mood and Anxiety Symptom Questionnaire - 30-item version) is a self-report questionnaire designed to measure symptoms of depression and anxiety. It separate symptoms that are shared between depression and anxiety from those that are more specific to each condition. The MASQ-30 includes 30 questions, divided into three main areas: Anhedonic Depression, which looks at symptoms like loss of interest or pleasure; Anxious Arousal, which focuses on physical signs of anxiety such as restlessness or a racing heart; and General Distress, which captures overall emotional discomfort common to both depression and anxiety. Each question asks how much the person has experienced a particular symptom in the past week, using a scale from 1 ("not at all") to 5 ("extremely").
Brain imaging | 8 weeks
  Non-invasive brain circuit quantification as assessed by functional magnetic resonance imaging metrics of activation and connectivity.
Cognitive-Emotional Behavioral Assessment | 8 weeks
  WebNeuro is a computerized cognitive-emotional behavioral assessment designed to objectively measure cognitive and emotional function.

SECONDARY OUTCOMES:
DARS: Dimensional Anhedonia Rating Scale | 8 weeks
  The DARS (Dimensional Anhedonia Rating Scale) is a brief, self-report tool developed to assess anhedonia, the reduced ability to experience pleasure-a key symptom in depression and other psychiatric disorders. It evaluates four domains of reward-related functioning: hobbies, food/drink, social activities, and sensory experiences (e.g., music, nature). For each domain, individuals rate items across several dimensions: interest, motivation, effort, and pleasure. Responses are given on a 5-point Likert scale, typically ranging from 0 to 4, with higher scores indicating greater engagement or enjoyment.
  The full scale includes 17 items, and the total score is calculated by summing the responses, with possible scores ranging from 0 to 68. Higher total scores reflect lower levels of anhedonia. Conversely, lower scores suggest greater anhedonia
PHQ-9: Patient Health Questionnaire-9 | 8 weeks
  The PHQ-9 (Patient Health Questionnaire-9) is a self-report screening tool designed to assess the presence and severity of depressive symptoms. It consists of 9 questions, each corresponding to one of the diagnostic criteria for major depressive disorder as outlined in the DSM. Respondents rate how often they have experienced each symptom over the past two weeks on a 4-point scale: 0 ("not at all"), 1 ("several days"), 2 ("more than half the days"), and 3 ("nearly every day"). The total score ranges from 0 to 27, with higher scores indicating more severe depressive symptoms. Scores are typically interpreted as follows: 0-4 (minimal depression), 5-9 (mild), 10-14 (moderate), 15-19 (moderately severe), and 20-27 (severe depression).
HAM-D-17: Hamilton Depression Rating Scale | 8 weeks
  The HAM-D-17 (Hamilton Depression Rating Scale), also known as the HDRS, is a clinician-administered assessment used to evaluate the severity of depressive symptoms in individuals diagnosed with depression. Each item is rated based on a structured interview, focusing on symptoms such as depressed mood, insomnia, anxiety, appetite disturbance, and suicidal ideation. Most items are scored on a scale from 0 to 4 or 0 to 2, depending on the symptom, with the total score ranging from 0 to 52 in the 17-item version. Interpretation of scores is generally as follows: 0-7 is considered normal or in remission, 8-13 indicates mild depression, 14-18 moderate, 19-22 severe, and 23 or higher very severe depression.
SWLS: Satisfaction With Life Scale | 8 weeks
  The Satisfaction With Life Scale (SWLS) is a brief, self-report questionnaire used to assess an individual's cognitive evaluation of life satisfaction. It consists of 5 items, each rated on a 7-point Likert scale ranging from 1 ("strongly disagree") to 7 ("strongly agree"), resulting in a total score ranging from 5 to 35. Higher scores indicate greater life satisfaction. The SWLS does not assess specific domains (e.g., health or work) but instead provides a broad measure of perceived well-being.
WHOQoL-BREF: The World Health Organization Quality of Life - BREF | 8 weeks
  The World Health Organization Quality of Life - BREF (WHOQOL-BREF) was developed by the World Health Organization to assess an individual's perceived quality of life. It includes 26 items that ask about a person's physical health, psychological well-being, social relationships, and environment. Each item is rated on a 5-point scale, with higher scores indicating a more positive perception of that area of life. The responses are grouped into four domain scores: Physical Health, Psychological Health, Social Relationships, and Environment. Scores for each domain are calculated and then transformed to a scale from 0 to 100, with higher scores reflecting better quality of life. The WHOQOL-BREF provides a broad yet efficient snapshot of how individuals feel about their overall well-being and daily functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sporn J, Ghaemi SN, Sambur MR, Rankin MA, Recht J, Sachs GS, Rosenbaum JF, Fava M. Pramipexole augmentation in the treatment of unipolar and bipolar depression: a retrospective chart review. Ann Clin Psychiatry. 2000 Sep;12(3):137-40. doi: 10.1023/a:1009060800999. PMID 10984002
- [Background] Goldberg JF, Burdick KE, Endick CJ. Preliminary randomized, double-blind, placebo-controlled trial of pramipexole added to mood stabilizers for treatment-resistant bipolar depression. Am J Psychiatry. 2004 Mar;161(3):564-6. doi: 10.1176/appi.ajp.161.3.564. PMID 14992985
- [Background] Lattanzi L, Dell'Osso L, Cassano P, Pini S, Rucci P, Houck PR, Gemignani A, Battistini G, Bassi A, Abelli M, Cassano GB. Pramipexole in treatment-resistant depression: a 16-week naturalistic study. Bipolar Disord. 2002 Oct;4(5):307-14. doi: 10.1034/j.1399-5618.2002.01171.x. PMID 12479663
- [Background] Inoue T, Kitaichi Y, Masui T, Nakagawa S, Boku S, Tanaka T, Suzuki K, Nakato Y, Usui R, Koyama T. Pramipexole for stage 2 treatment-resistant major depression: an open study. Prog Neuropsychopharmacol Biol Psychiatry. 2010 Dec 1;34(8):1446-9. doi: 10.1016/j.pnpbp.2010.07.035. Epub 2010 Aug 11. PMID 20708060
- [Background] Hori H, Kunugi H. The efficacy of pramipexole, a dopamine receptor agonist, as an adjunctive treatment in treatment-resistant depression: an open-label trial. ScientificWorldJournal. 2012;2012:372474. doi: 10.1100/2012/372474. Epub 2012 Aug 1. PMID 22919308
- [Background] Dell'Osso B, Ketter TA. Assessing efficacy/effectiveness and safety/tolerability profiles of adjunctive pramipexole in bipolar depression: acute versus long-term data. Int Clin Psychopharmacol. 2013 Nov;28(6):297-304. doi: 10.1097/YIC.0b013e3283639015. PMID 24081199
- [Background] Strejilevich SA, Martino DJ, Igoa A, Manes F. Pathological gambling in a bipolar patient treated with pramipexole. J Neuropsychiatry Clin Neurosci. 2011 Winter;23(1):E2-3. doi: 10.1176/jnp.23.1.jnpe2. No abstract available. PMID 21304118
- [Background] El-Mallakh RS, Penagaluri P, Kantamneni A, Gao Y, Roberts RJ. Long-term use of pramipexole in bipolar depression: a naturalistic retrospective chart review. Psychiatr Q. 2010 Sep;81(3):207-13. doi: 10.1007/s11126-010-9130-6. PMID 20425143
- [Background] Cassano P, Lattanzi L, Soldani F, Navari S, Battistini G, Gemignani A, Cassano GB. Pramipexole in treatment-resistant depression: an extended follow-up. Depress Anxiety. 2004;20(3):131-8. doi: 10.1002/da.20038. PMID 15549689
- [Background] Takahashi M, Nishida S, Nakamura M, Kobayashi M, Matsui K, Ito E, Usui A, Inoue Y. Restless legs syndrome augmentation among Japanese patients receiving pramipexole therapy: Rate and risk factors in a retrospective study. PLoS One. 2017 Mar 6;12(3):e0173535. doi: 10.1371/journal.pone.0173535. eCollection 2017. PMID 28264052
- [Background] Perugi G, Toni C, Ruffolo G, Frare F, Akiskal H. Adjunctive dopamine agonists in treatment-resistant bipolar II depression: an open case series. Pharmacopsychiatry. 2001 Jul;34(4):137-41. doi: 10.1055/s-2001-15872. PMID 11518474
- [Background] Aiken CB. Pramipexole in psychiatry: a systematic review of the literature. J Clin Psychiatry. 2007 Aug;68(8):1230-6. PMID 17854248
- [Background] Zarate CA Jr, Payne JL, Singh J, Quiroz JA, Luckenbaugh DA, Denicoff KD, Charney DS, Manji HK. Pramipexole for bipolar II depression: a placebo-controlled proof of concept study. Biol Psychiatry. 2004 Jul 1;56(1):54-60. doi: 10.1016/j.biopsych.2004.03.013. PMID 15219473
- [Background] Corrigan MH, Denahan AQ, Wright CE, Ragual RJ, Evans DL. Comparison of pramipexole, fluoxetine, and placebo in patients with major depression. Depress Anxiety. 2000;11(2):58-65. doi: 10.1002/(sici)1520-6394(2000)11:23.0.co;2-h. PMID 10812530
- [Background] Chaudhuri KR, Rizos A, Sethi KD. Motor and nonmotor complications in Parkinson's disease: an argument for continuous drug delivery? J Neural Transm (Vienna). 2013 Sep;120(9):1305-20. doi: 10.1007/s00702-013-0981-5. Epub 2013 Mar 2. PMID 23456290
- [Background] Drijgers RL, Verhey FR, Tissingh G, van Domburg PH, Aalten P, Leentjens AF. The role of the dopaminergic system in mood, motivation and cognition in Parkinson's disease: a double blind randomized placebo-controlled experimental challenge with pramipexole and methylphenidate. J Neurol Sci. 2012 Sep 15;320(1-2):121-6. doi: 10.1016/j.jns.2012.07.015. Epub 2012 Jul 22. PMID 22824349
- [Background] Miura S, Kida H, Nakajima J, Noda K, Nagasato K, Ayabe M, Aizawa H, Hauser M, Taniwaki T. Anhedonia in Japanese patients with Parkinson's disease: analysis using the Snaith-Hamilton Pleasure Scale. Clin Neurol Neurosurg. 2012 May;114(4):352-5. doi: 10.1016/j.clineuro.2011.11.008. Epub 2011 Dec 2. PMID 22137783
- [Background] Fujiwara S, Kimura F, Hosokawa T, Ishida S, Sugino M, Hanafusa T. Anhedonia in Japanese patients with Parkinson's disease. Geriatr Gerontol Int. 2011 Jul;11(3):275-81. doi: 10.1111/j.1447-0594.2010.00678.x. Epub 2011 Jan 17. PMID 21241445
- [Background] Hamidovic A, Kang UJ, de Wit H. Effects of low to moderate acute doses of pramipexole on impulsivity and cognition in healthy volunteers. J Clin Psychopharmacol. 2008 Feb;28(1):45-51. doi: 10.1097/jcp.0b013e3181602fab. PMID 18204340
- [Background] Lemke MR, Brecht HM, Koester J, Kraus PH, Reichmann H. Anhedonia, depression, and motor functioning in Parkinson's disease during treatment with pramipexole. J Neuropsychiatry Clin Neurosci. 2005 Spring;17(2):214-20. doi: 10.1176/jnp.17.2.214. PMID 15939976
- [Background] Reichmann H, Brecht MH, Koster J, Kraus PH, Lemke MR. Pramipexole in routine clinical practice: a prospective observational trial in Parkinson's disease. CNS Drugs. 2003;17(13):965-73. doi: 10.2165/00023210-200317130-00003. PMID 14533946
- [Background] Fawcett J, Rush AJ, Vukelich J, Diaz SH, Dunklee L, Romo P, Yarns BC, Escalona R. Clinical Experience With High-Dosage Pramipexole in Patients With Treatment-Resistant Depressive Episodes in Unipolar and Bipolar Depression. Am J Psychiatry. 2016 Feb 1;173(2):107-11. doi: 10.1176/appi.ajp.2015.15060788. No abstract available. PMID 26844792